CLINICAL TRIAL: NCT05802615
Title: Protective Assets Reinforced With Integrated Care and TechnologY (PARITY) Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0076-23-EP
Record Dates: First submitted 2023-03-19; First posted 2023-04-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2024-12

CONDITIONS: Maternal Health; Blood Pressure
MeSH Terms: interventions — Parity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARITY (Experimental): Participants will take part in the Protective Assets Reinforced with Integrated care and TechnologY (PARITY) program which is community-based doula support, community resources, and a mobile technology platform that reinforces individual strengths through positive messaging and by promoting wellness (sleep, physical activity, nutrition, prenatal care adherence) in Black pregnant women.
  Interventions: Behavioral: PARITY; Other: Usual Care
- Control (Placebo Comparator): Participants will obtain prenatal care from their usual care provider and a handout on healthy pregnancy.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: PARITY — The PARITY program reinforces strengths through consistent, community-based Black doula support and protective asset (personal strengths) focused messaging. PARITY promotes wellness-related behaviors (nutrition, physical activity, sleep, and healthcare adherence) and promotes and builds empowered strengths (self-efficacy, social support, motivation, resilience, problem-solving, and self-regulation) through mobile technology and doula support.
  Arms: PARITY
Other: Usual Care — Participants will obtain prenatal care from their usual care provider and a handout on healthy pregnancy.

SUMMARY:
This study will determine the feasibility and acceptability of the Protective Assets Reinforced with Integrated care and TechnologY (PARITY) program, to test the clinical, behavioral, and strength building efficacy of the PARITY program and explore how it achieves its outcomes in pregnant Black women. PARITY is a program that provides community-based doula support, community resources, and a mobile technology platform that reinforces individual strengths (referred to as protective assets) through positive messaging and by promoting wellness.

DETAILED DESCRIPTION:
The overall objective of this study is to determine the feasibility and acceptability of the Protective Assets Reinforced with Integrated care and TechnologY (PARITY) program, to test the clinical, behavioral, and strength building efficacy of the PARITY program and explore how it achieves its outcomes in pregnant Black women. PARITY is a program that provides community-based doula support, community resources, and a mobile technology platform that reinforces individual strengths (referred to as protective assets) through positive messaging and by promoting wellness (sleep, physical activity, nutrition, prenatal care adherence) in Black pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Black race
* Pregnant with gestational age 20-28 weeks at enrollment
* Ability to read and write in English language
* Planning to give birth at a healthcare facility & receive obstetrical care with a healthcare record
* Reside within 20 minutes of the Lincoln/Omaha, NE metro area
* Owns a smartphone with internet access

Exclusion Criteria:

-

Ages: 19 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be pregnant females
Enrollment: 60 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Maternal Blood Pressure | 20 weeks
  Participant blood pressure (systolic and diastolic) (continuous) as well as blood pressure classifications hypertension (>140/90); Severe hypertension (>160/110).
Maternal Blood Pressure | 36 weeks
  Participant blood pressure (systolic and diastolic) (continuous) as well as blood pressure classifications hypertension (>140/90); Severe hypertension (>160/110).
Maternal Blood Pressure | Birth (approximately 36-42 weeks)
  Participant blood pressure (systolic and diastolic) (continuous) as well as blood pressure classifications hypertension (>140/90); Severe hypertension (>160/110).
Maternal Blood Pressure | 6-12 weeks postpartum
  Participant blood pressure (systolic and diastolic) (continuous) as well as blood pressure classifications hypertension (>140/90); Severe hypertension (>160/110).
Feasibility, Enrollment | Baseline
  Percentage of eligible individuals who agree to participate in the trial
Feasibility, Attrition | Completion of Study (~24 months)
  Percentage of eligible individuals who complete the data
Feasibility, Adherence | Completion of Study (~24 months)
  Number of intervention sessions completed by study participants

SECONDARY OUTCOMES:
Gestational Weight Gain | 20 weeks, 36 weeks, Birth, 6 weeks postpartum.
  Amount of weight gained in pounds
Delivery Modality | Birth (approximately 36-42 weeks)
  Modality of birth (Vaginal, Cesarean, Assisted Vaginal delivery)

OTHER OUTCOMES:
Nutritional Intake | Baseline, 6-12 weeks postpartum
  Nutritional intake will be measured with the Multifactor Screener, 2000 as used in the Observing Protein and Energy Nutrition (OPEN) Study. This instrument measures approximate intakes of fruits and vegetables, percentage energy from fat, and fiber. Respondents report how frequently they consume foods in 16 categories and type of milk consumed.
Physical Activity | Baseline, 6-12 weeks postpartum
  Physical activity will be measured with the International Physical Activity Questionnaire short-form (IPAQ-SF). The IPAQ-SF consists of 9 items and provides information on the time spent walking, in vigorous and moderate intensity activity and in sedentary activity.
Sleep quality | Baseline, 6-12 weeks postpartum
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI. The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score.
Healthcare Adherence | Pregnancy continuum, measured at 12 weeks postpartum retrospectively via the medical record
  Healthcare adherence will be measured by number of healthcare appointments measured in the medical record.
Self-efficacy | Baseline, 6-12 weeks postpartum
  Self-efficacy will be measured using the GSE General Self Efficacy (GSE) Scale: The GSE is a one-dimensional self-report measure that features a 10-item questionnaire assessing the optimistic self-beliefs of individuals to cope with a variety of difficult demands in life. The response options are presented along a 4-point Likert scale for each item.
Social support | Baseline, 6-12 weeks postpartum
  Social support will be measured with the 10 item Social Provisions Scale (SPS-10). The SPS-10 assesses five forms of social provisions: attachment, guidance, social integration, reliable alliance, and reassurance of worth. Each item is rated on a four-point Likert scale.
Problem-solving | Baseline, 6-12 weeks postpartum
  Problem solving will be measured with the Problem-Solving Inventory (PSI). The PSI measures how well individuals make decisions and their problem-solving abilities. The PSI includes 32 items using a 6-point Likert scale.
Motivation | Baseline, 6-12 weeks postpartum
  Motivation will be measured with the Self-Motivation Inventory (SMI). The SMI is a 40 item 5 point Likert scale.
Resilience | Baseline, 6-12 weeks postpartum
  Resilience will be measured using the 10 item Connor-Davidson Resilience Scale (CD-RISC 10). The CD-RISC 10 a unidimensional self-reported scale consisting of 10-items measuring resilience. Respondents rate items on a 5-point Likert scale.
Self-Regulation | Baseline, 6-12 weeks postpartum
  Self-Regulation will be measured with the index of self-regulation (ISR). The ISR is a nine-item scale that measures level of self-regulation for health behavior change. Respondents rate items on a 5-point Likert scale.
Discrimination | Baseline, 6-12 weeks postpartum
  Discrimination will be measured using the Everyday Discrimination Scale (EDS). The EDS measures frequency of chronic and routine unfair treatment in everyday life. Respondents are asked to report how often they experience unfair treatment in their day-to-day life on a 6-point Likert scale.
Neighborhood | Baseline
  Neighborhood will be assessed using the Neighborhood Collective Efficacy - Community Cohesion and Informal Social Control protocol. This protocol includes 10 Likert-style questions from the Project on Human Development in Chicago Neighborhoods (PHDCN). The Social Cohesion and Informal Social Control subscales include five items each.
Acceptability and Experience | 12 weeks postpartum
  Select intervention participants only (10-15). Qualitative interview to discuss acceptability and experience with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Mollard, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mollard E, Cooper Owens D, Bach C, Gaines C, Maloney S, Moore T, Wichman C, Shah N, Balas M. Protective Assets Reinforced With Integrated Care and Technology (PARITY): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Aug 8;13:e58580. doi: 10.2196/58580. PMID 39116423